CLINICAL TRIAL: NCT04507503
Title: An Open-Label Expanded Access Program of Futibatinib (TAS-120) In Patients With Advanced Cholangiocarcinoma Harboring FGFR2 Gene Rearrangements
Brief Title: Expanded Access Study of TAS-120 in Patients With Advanced Cholangiocarcinoma Harboring FGFR2 Gene Rearrangements
Status: Approved for marketing | Type: Expanded Access
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TAS-120-401
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Advanced Cholangiocarcinoma
Keywords: Cholangiocarcinoma; CCA; FGFR2 Gene Rearrangements; TAS-120; Futibatinib
MeSH Terms: conditions — Cholangiocarcinoma | interventions — futibatinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: TAS-120 — Futibatinib 20mg QD orally on a 28 days cycle
  Other Names: Futibatinib

SUMMARY:
The objective of the study is to provide access to TAS-120 to patients With Advanced Cholangiocarcinoma Harboring FGFR2 Gene Rearrangements.

DETAILED DESCRIPTION:
This is an open-label study to provide expanded access to TAS-120 prior to its commercial availability for patients with Advanced Cholangiocarcinoma Harboring FGFR2 Gene Rearrangements who have failed standard therapy or who are unable to tolerate standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. >18 years of age.
3. Histologically confirmed, locally advanced, or metastatic, or recurrent unresectable CCA harboring FGFR2 gene rearrangements based on testing performed by a qualified (CLIA-certified) laboratory.
4. Patient has failed standard therapy or standard therapy is not tolerated.
5. Has measurable or non-measurable lesion(s).
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Adequate organ function.

Exclusion Criteria:

1. History and/or current evidence of non-tumor related alteration of calcium-phosphorus homeostasis.
2. History and/or current evidence of clinically significant ectopic mineralization/calcification.
3. History and/or current evidence of clinically significant retinal disorder confirmed by retinal examination.
4. A serious illness or medical condition(s)
5. Pregnant or breast-feeding female

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Banner MD Anderson, Gilbert, Arizona
  - University of California, San Francisco (UCSF), San Francisco, California
  - UCLA Division of Hematology-Oncology, Santa Monica, California
  - Mount Sinai Center of Florida, Miami Beach, Florida
  - Advent Health Orlando, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Kansas Cancer Center, Lee's Summit, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - MD Anderson, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Aurora Cancer care, Grafton, Wisconsin